CLINICAL TRIAL: NCT07358546
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Pharmacokinetics and Safety of Efimosfermin Alfa in Adults With Varying Degrees of Hepatic Impairment Due to Steatotic Liver Disease
Brief Title: A Study of Efimosfermin Alfa in Adults With Hepatic Impairment
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 306836
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: efimosfermin alfa; Alcohol; Hepatic Impairment; Steatotic liver disease; Metabolic Dysfunction-Associated Steatohepatitis; Pharmacokinetics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Masking Description: open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efimosfermin alfa in participants with moderate hepatic impairment due to MASH without alcohol (Experimental): All participants will receive efimosfermin alfa. Participants will have moderate hepatic impairment (Child-Pugh B) due to Metabolic Dysfunction-Associated Steatohepatitis (MASH) with typical average daily alcohol consumption threshold of less than or equal to (<=) 30 gram ethanol or <=5 standard drinks (men), or <=16 gram ethanol or <=4 standard drinks (women) per day for 3 months prior to Screening.
  Interventions: Drug: Efimosfermin alfa
- Efimosfermin alfa in participants with moderate hepatic impairment due to MASH with alcohol (Experimental): All participants will receive efimosfermin alfa. Participants will have moderate hepatic impairment (Child-Pugh B) due to MASH with typical average daily alcohol consumption threshold of greater than (>) 30 gram ethanol or >5 standard drinks (men) or >16 gram ethanol or >4 standard drinks (women) per day for 3 months prior to Screening.
  Interventions: Drug: Efimosfermin alfa
- Efimosfermin alfa in participants with severe hepatic impairment due to MASH despite of alcohol use (Experimental): All participants will receive efimosfermin alfa. Participants will have severe hepatic impairment (Child-Pugh C) due to MASH with any typical daily alcohol consumption.
  Interventions: Drug: Efimosfermin alfa

INTERVENTIONS:
Drug: Efimosfermin alfa — Efimosfermin alfa to be administrated subcutaneously

SUMMARY:
This study is designed to study the pharmacokinetic (PK) and safety profiles of a single dose of efimosfermin alfa in participants with varying degrees of Hepatic Impairment (HI) (assessed by Child-Pugh score) due to steatotic liver disease, with and without significant alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 years and 70 years of age inclusive
* Body Mass Index (BMI) within the range 23 - 40 kilogram per square meter (kg/m^2)
* Male or female participants
* Participant has liver cirrhosis with a grade of hepatic impairment that can be classified as a discrete Child-Pugh class. Participants must:

  * Have a clinical diagnosis of liver cirrhosis in the participant's medical history corroborated by previous liver biopsy, medical imaging or compatible biochemical profile, and
  * Be classed during screening as one of the following Child-Pugh classes:

    * Child-Pugh B: Score 7-9 or
    * Child-Pugh C: Score 10-15
* Chronic (>6 months) HI which is currently stable (no acute episodes of illness within the previous 1 month prior to Screening (Visit 1) due to deterioration in hepatic function). Participants must also remain stable throughout the Screening period. Assessment of the stability of the participant's hepatic function will be determined by the investigator.

Exclusion Criteria:

* History of extrahepatic disorders possibly related to etiology of cirrhosis.
* History of cryoglobulinemia.
* Participants with Grade 3
* Participants with refractory encephalopathy or significant central nervous system disease
* History of gastric or esophageal variceal bleeding within the past 6 months and for which varices have not been adequately
* Other primary causes of liver disease Steatotic liver disease must be the primary cause of liver disease.
* Clinically significant abnormalities affecting physical health in medical history, or on physical examination, that could interfere with or for which treatment could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study
* Current, or history of known hepatocellular carcinoma (HCC).
* Participants with transjugular intrahepatic portosystemic shunt (TIPS) placement.
* Presence of hepatopulmonary or hepatorenal syndrome.
* Presence of primarily cholestatic liver diseases.
* Evidence of symptomatic or complicated cholecystitis of
* History of pancreatic injury, pancreatitis, or other pancreatic disease.
* History of liver transplantation.
* Participants with signs of active infection
* History of adrenal gland disease or using treatment that affects the hypothalamic-pituitary-adrenal axis.
* History of significant bone disease such as osteoporosis
* Psychosocial features that, in the opinion of the investigator, increase the likelihood of loss to follow-
* History or presence of drug abuse.
* Use of other investigational drugs at the time of screening, or within 5 half-lives or 30 days prior to study intervention, whichever was longer; or longer if required by local regulations
* Have previously taken efimosfermin alfa
* Participants with Alanine Aminotransferase (ALT) value >3 x upper limit of normal (ULN)
* Average of triplicate corrected QT interval, (QTc) >480 msec in (for male and female participants)participants with bundle branch block at Day -1 (Visit 2) (a mean of triplicate measurements should be used to confirm that the participant meets exclusion criterion).
* For participants in the MASH with alcohol category, significant risk of withdrawal symptoms:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Area under the serum drug concentration versus time curve from time zero to infinity (AUC[0-inf]) of efimosfermin alfa | Up to 90 Days
Maximum observed serum drug concentration (Cmax) of efimosfermin alfa | Up to 90 Days

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs), treatment related AEs and serious adverse events (SAEs) | Up to 90 Days
Number of participants with Clinically significant changes in hematology, chemistry, and urinalysis parameters | Up to 90 Days
Number of participants with Clinically significant changes in Vital signs and 12-lead electrocardiogram (ECG) findings | Up to 90 Days
Area under the serum drug concentration versus time curve from time zero to the time of the last quantifiable concentration (AUC[0-t]) of efimosfermin alfa | Up to 90 Days
Time to maximum observed serum drug concentration (Tmax) of efimosfermin alfa | Up to 90 Days
Apparent terminal phase half-life (t1/2) of efimosfermin alfa | Up to 90 Days
Time prior to the first measurable (non-zero) serum concentration (Tlag) of efimosfermin alfa | Up to 90 Days
Apparent clearance (CL/F) of efimosfermin alfa | Up to 90 days
Apparent terminal phase volume of distribution (Vz/F) of efimosfermin alfa | Up to 90 days
Terminal elimination rate constant (Lambda z) of efimosfermin alfa | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf